CLINICAL TRIAL: NCT06876012
Title: Impact of Tai Chi on Balance and Fall Risk in Patients With Cervical Myelopathy
Brief Title: Impact of Tai Chi in Cervical Myelopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Scott Daffner, Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2409042637
Record Dates: First submitted 2025-03-12; First posted 2025-03-14 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cervical Myelopathy; Balance Assessment; Fall Risk
Keywords: Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Control) (No Intervention): Subjects will follow the current standard of care procedures utilized by the WVU Spine Center.
- Intervention Group (Tai Chi) (Experimental): These subjects will participate in 12 sessions of Tai Chi class over the course of 6 weeks.
  Interventions: Other: Tai Chi Program

INTERVENTIONS:
Other: Tai Chi Program — Twelve sessions (six weeks) of a Tai Chi Program to assist with balance and fall risk.
  Arms: Intervention Group (Tai Chi)

SUMMARY:
The goal of this observational study is to determine if patients with cervical myelopathy who participate in a Tai Chi program will demonstrate improved gait and balance compared to patients who undergo usual care.

Participants must be 18 years or older and have a diagnosis of cervical myelopathy.

DETAILED DESCRIPTION:
Patients who meet inclusion criteria and choose to participate will be randomized to either participate in a Tai Chi falls-prevention program or continue with usual care. Those in the Tai Chi program will attend a pre-determined number of Tai Chi classes for a period of approximately 6-8 weeks. Investigators will assess their gait and balance at the time of enrollment and at several timepoints after they have participated in the class (similar timepoints for those randomized to usual care).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cervical Myelopathy with planned surgery
* 18 years of age or older
* Able to participate in intervention (attend and participate in classes)

Exclusion Criteria:

* Wheelchair bound at initial visit
* Other verified potential cause of gait instability/balance problems
* Unable to participate in intervention (unable to attend/participate in classes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test - Baseline | Baseline
  Establish a baseline score. The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults.
  Setup: The person sits in a standard armchair. Instructions: On the command "Go," the person stands up, walks 3 meters (about 10 feet) at a comfortable pace, turns around, walks back to the chair, and sits down.
  Timing: The time taken from the command "Go" until the person sits back down is recorded. This is recorded in minutes:seconds.
  Scoring Normal Mobility: Completing the test in less than 10 seconds. Mild Mobility Impairment: Completing the test in 10-19 seconds. Moderate Mobility Impairment: Completing the test in 20-29 seconds. Severe Mobility Impairment: Taking 30 seconds or more to complete the test. A time of 12 seconds or more indicates a higher risk of falling.
Timed Up and Go Test - 6 weeks | 6 weeks post-operatively
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults. This is recorded in minutes:seconds.
  Setup: The person sits in a standard armchair. Instructions: On the command "Go," the person stands up, walks 3 meters (about 10 feet) at a comfortable pace, turns around, walks back to the chair, and sits down.
  Timing: The time taken from the command "Go" until the person sits back down is recorded. This is recorded in minutes:seconds.
  Scoring Normal Mobility: Completing the test in less than 10 seconds. Mild Mobility Impairment: Completing the test in 10-19 seconds. Moderate Mobility Impairment: Completing the test in 20-29 seconds. Severe Mobility Impairment: Taking 30 seconds or more to complete the test. A time of 12 seconds or more indicates a higher risk of falling.
Timed Up and Go Test - 3 months | 3 months post-operatively
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults. This is recorded in minutes:seconds.
  Setup: The person sits in a standard armchair. Instructions: On the command "Go," the person stands up, walks 3 meters (about 10 feet) at a comfortable pace, turns around, walks back to the chair, and sits down.
  Timing: The time taken from the command "Go" until the person sits back down is recorded. This is recorded in minutes:seconds.
  Scoring Normal Mobility: Completing the test in less than 10 seconds. Mild Mobility Impairment: Completing the test in 10-19 seconds. Moderate Mobility Impairment: Completing the test in 20-29 seconds. Severe Mobility Impairment: Taking 30 seconds or more to complete the test. A time of 12 seconds or more indicates a higher risk of falling.
Timed Up and Go Test - 6 months | 6 months post-operatively
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults. This is recorded in minutes:seconds.
  Setup: The person sits in a standard armchair. Instructions: On the command "Go," the person stands up, walks 3 meters (about 10 feet) at a comfortable pace, turns around, walks back to the chair, and sits down.
  Timing: The time taken from the command "Go" until the person sits back down is recorded. This is recorded in minutes:seconds.
  Scoring Normal Mobility: Completing the test in less than 10 seconds. Mild Mobility Impairment: Completing the test in 10-19 seconds. Moderate Mobility Impairment: Completing the test in 20-29 seconds. Severe Mobility Impairment: Taking 30 seconds or more to complete the test. A time of 12 seconds or more indicates a higher risk of falling.
Timed Up and Go Test - 12 months | 12 months post-operatively
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults. This is recorded in minutes:seconds.
  Setup: The person sits in a standard armchair. Instructions: On the command "Go," the person stands up, walks 3 meters (about 10 feet) at a comfortable pace, turns around, walks back to the chair, and sits down.
  Timing: The time taken from the command "Go" until the person sits back down is recorded. This is recorded in minutes:seconds.
  Scoring Normal Mobility: Completing the test in less than 10 seconds. Mild Mobility Impairment: Completing the test in 10-19 seconds. Moderate Mobility Impairment: Completing the test in 20-29 seconds. Severe Mobility Impairment: Taking 30 seconds or more to complete the test. A time of 12 seconds or more indicates a higher risk of falling.

SECONDARY OUTCOMES:
10-Step Tandem Gait Test - Baseline | Baseline
  Establish a baseline score. The 10-Step Tandem Gait Test asks participants to walk a straight line making a toe-to-heal touch with each step at the subject's own velocity. The number of steps made before the first misstep is counted. After first 10-step tandem gait test, the subject turns around and repeats the tandem gait test in the same line and the number of steps is counted in the same manner. This is a graded score from 0-4. The higher grade demonstrates better gait.
  Scoring Grade 4: Completes all 10 steps without any instability. Grade 3: Completes 8-9 steps with minimal instability. Grade 2: Completes 6-7 steps with moderate instability. Grade 1: Completes 4-5 steps with significant instability. Grade 0: Completes fewer than 4 steps or is unable to perform the test due to severe instability.
10-Step Tandem Gait Test - 6 weeks | 6 weeks post-operatively
  The 10-Step Tandem Gait Test asks participants to walk a straight line making a toe-to-heal touch with each step at the subject's own velocity. The number of steps made before the first misstep is counted. After first 10-step tandem gait test, the subject turns around and repeats the tandem gait test in the same line and the number of steps is counted in the same manner. This is a graded score from 0-4. The higher grade demonstrates better gait.
  Scoring Grade 4: Completes all 10 steps without any instability. Grade 3: Completes 8-9 steps with minimal instability. Grade 2: Completes 6-7 steps with moderate instability. Grade 1: Completes 4-5 steps with significant instability. Grade 0: Completes fewer than 4 steps or is unable to perform the test due to severe instability.
10-Step Tandem Gait Test - 3 months | 3 months post-operatively
  The 10-Step Tandem Gait Test asks participants to walk a straight line making a toe-to-heal touch with each step at the subject's own velocity. The number of steps made before the first misstep is counted. After first 10-step tandem gait test, the subject turns around and repeats the tandem gait test in the same line and the number of steps is counted in the same manner. This is a graded score from 0-4. The higher grade demonstrates better gait.
  Scoring Grade 4: Completes all 10 steps without any instability. Grade 3: Completes 8-9 steps with minimal instability. Grade 2: Completes 6-7 steps with moderate instability. Grade 1: Completes 4-5 steps with significant instability. Grade 0: Completes fewer than 4 steps or is unable to perform the test due to severe instability.
10-Step Tandem Gait Test - 6 months | 6 months post-operatively
  The 10-Step Tandem Gait Test asks participants to walk a straight line making a toe-to-heal touch with each step at the subject's own velocity. The number of steps made before the first misstep is counted. After first 10-step tandem gait test, the subject turns around and repeats the tandem gait test in the same line and the number of steps is counted in the same manner. This is a graded score from 0-4. The higher grade demonstrates better gait.
  Scoring Grade 4: Completes all 10 steps without any instability. Grade 3: Completes 8-9 steps with minimal instability. Grade 2: Completes 6-7 steps with moderate instability. Grade 1: Completes 4-5 steps with significant instability. Grade 0: Completes fewer than 4 steps or is unable to perform the test due to severe instability.
10-Step Tandem Gait Test - 12 Month | 12 months post-operatively
  The 10-Step Tandem Gait Test asks participants to walk a straight line making a toe-to-heal touch with each step at the subject's own velocity. The number of steps made before the first misstep is counted. After first 10-step tandem gait test, the subject turns around and repeats the tandem gait test in the same line and the number of steps is counted in the same manner. This is a graded score from 0-4. The higher grade demonstrates better gait.
  Scoring Grade 4: Completes all 10 steps without any instability. Grade 3: Completes 8-9 steps with minimal instability. Grade 2: Completes 6-7 steps with moderate instability. Grade 1: Completes 4-5 steps with significant instability. Grade 0: Completes fewer than 4 steps or is unable to perform the test due to severe instability.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Daffner, MD, Principal Investigator — West Virginia University School of Medicine, Department of Orthopaedics; Andrya Durr, PhD, Study Director — West Virginia University School of Public Health

REFERENCES:
- [Background] Chen Y, Wan A, Mao M, Sun W, Song Q, Mao D. Tai Chi practice enables prefrontal cortex bilateral activation and gait performance prioritization during dual-task negotiating obstacle in older adults. Front Aging Neurosci. 2022 Nov 18;14:1000427. doi: 10.3389/fnagi.2022.1000427. eCollection 2022. PMID 36466597
- [Background] Zu Y, Luo L, Chen X, Xie H, Yang CR, Qi Y, Niu W. Characteristics of corticomuscular coupling during wheelchair Tai Chi in patients with spinal cord injury. J Neuroeng Rehabil. 2023 Jun 17;20(1):79. doi: 10.1186/s12984-023-01203-x. PMID 37330516
- [Background] Tsang WW, Gao KL, Chan KM, Purves S, Macfarlane DJ, Fong SS. Sitting tai chi improves the balance control and muscle strength of community-dwelling persons with spinal cord injuries: a pilot study. Evid Based Complement Alternat Med. 2015;2015:523852. doi: 10.1155/2015/523852. Epub 2015 Jan 21. PMID 25688276
- [Background] Qi Y, Zhang X, Zhao Y, Xie H, Shen X, Niu W, Wang Y. The effect of wheelchair Tai Chi on balance control and quality of life among survivors of spinal cord injuries: A randomized controlled trial. Complement Ther Clin Pract. 2018 Nov;33:7-11. doi: 10.1016/j.ctcp.2018.07.004. Epub 2018 Jul 20. PMID 30396629
- [Background] Chen W, Li M, Li H, Lin Y, Feng Z. Tai Chi for fall prevention and balance improvement in older adults: a systematic review and meta-analysis of randomized controlled trials. Front Public Health. 2023 Sep 1;11:1236050. doi: 10.3389/fpubh.2023.1236050. eCollection 2023. PMID 37736087
- [Background] Voukelatos A, Cumming RG, Lord SR, Rissel C. A randomized, controlled trial of tai chi for the prevention of falls: the Central Sydney tai chi trial. J Am Geriatr Soc. 2007 Aug;55(8):1185-91. doi: 10.1111/j.1532-5415.2007.01244.x. PMID 17661956